CLINICAL TRIAL: NCT02900118
Title: Imaging Evaluation of the Therapeutic Response of Breast Cancer Bone Metastasis
Brief Title: Imaging Evaluation of the Therapeutic Response of Breast Cancer Bone Metastasis (EMOS)
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: EMOS-1207
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Bone metastasis; PET-CT; whole-body MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients with breast cancer bone metastasis at the initial diagnosis.
- Group 2: Patients with breast cancer bone metastasis in a metastatic bone relapse.
- Group 3: Patients with breast cancer bone metastasis with a progression of bone metastasis.

SUMMARY:
Breast cancers are among the cancers that metastasize the most to the skeleton. The appearance of bone metastasis, whether they are initials or during a relapse, is a turning point of the disease, due to the additional morbidity they imply (pain, pathologic fractures, hypercalcaemia, neurological compression, etc.). A specific treatment of these metastasis is often undertaken, usually a chemotherapy or hormone therapy. It is important to evaluate the efficacy of this treatment in order to know whether to continue or change it depending on the response observed. But there is no consensus at this time on paraclinical examinations enabling this monitoring. Also, if some criteria for assessing bone metastasis in imaging and nuclear medicine (MDA, PERCIST, EORTC) have been published in the literature, none is formally validated and evaluation in routine practice remains subjective.

The main objective of our study is to determine if the PET-CT and the whole-body MRI are in agreement on the status of bone metastasis (stability, progression, partial response, complete response).

DETAILED DESCRIPTION:
The oncologist includes patients responding to criteria and not opposing the collection of their data. He submits a request for whole-body MRI and PET-CT to the Medical Imaging and Nuclear Medicine departments of the Oscar Lambret Centre. If the patient has benefited within the previous 15 days of any of these examinations, it is not performed again : it will serve as an initial examination. Following these examinations, the oncologist completes the reading grid. A clinical examination and a questioning with the main stages of the disease is performed and data are reported in the dedicated sheet. A prescription of tumor markers and of bone remodeling is performed (in the absence of recent results), and the results are reported on the same sheet.

After 3 cycles (of intravenous chemotherapy) or 3 months of hormone therapy, the oncologist submits a new request for whole-body MRI and PET-CT. The MRI and PET-CT should conclude to a status : progression, stability, partial response, complete response. The reading grid is completed again. MDA criteria (MRI and PET-CT), PERCIST and EORTC (PET-CT only) are determined. Target lesions (1 to 3) are defined for each examination and a measure of the ADC and the SUV is performed for each lesion on the initial and follow-up examinations.

After these examinations, the patient is reviewed by his oncologist for a new clinical examination, the announcement of the status of bone metastasis and the possible adaptation of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with breast cancer bone metastasis :

   * at the initial diagnosis (group 1).
   * in a metastatic bone relapse (group 2).
   * with a progression of bone metastasis (group 3).
2. Treatment (hormone therapy, chemotherapy) not undertaken (group 1) or prior therapeutic change (group 2 and 3).
3. Patient not opposing the use of its data.

Exclusion Criteria:

1. Claustrophobic patient
2. Patient with an uncontrolled diabetes (fasting glucose < 1.6 g / l)
3. Patient with a pace-maker or another material incompatible with the MRI 3 Tesla
4. Very algetic patient (Visual Analog Scale (VAS) > 7)
5. Pregnant or breastfeeding women
6. Patient under 18 or under guardianship
7. Movement disorders (Parkinson disease, etc.) or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included are patients seen in consultation for discovery or monitoring of breast cancer bone metastasis at the Oscar Lambret Centre, who meet the eligibility criteria and who have given their consent.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the therapeutic response. | Cycle 3 (each cycle is 28 days)

SECONDARY OUTCOMES:
Evaluation of the concordance of the Apparent Diffusion Coefficient (ADC) and the Standardized Uptake Value (SUV). | At baseline
Evaluation of the concordance of the Apparent Diffusion Coefficient (ADC) and the Standardized Uptake Value (SUV). | Cycle 3 (each cycle is 28 days)
Evaluation of the consistency in the detection of lesions. | Cycle 3 (each cycle is 28 days)
Evaluation of the criteria PERCIST (PET Response Criteria in Solid Tumors) | Cycle 3 (each cycle is 28 days)
Evaluation of the criteria MDA (Minimal Disease Activity) | Cycle 3 (each cycle is 28 days)
Evaluation of the criteria EORTC (European Organisation for Research and Treatment of Cancer). | Cycle 3 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Armelle RENAUD, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No